CLINICAL TRIAL: NCT04878705
Title: A Randomized, Double-blind, Placebo-controlled, Single Dose, Escalation, Phase I Clinical Trial to Evaluate the Safety and Tolerability of TWP-201 in Healthy Female Subjects
Brief Title: Safety and Tolerability of TWP-201 in Healthy Female Subjects
Status: Unknown | Phase: Phase 1 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Shandong TheraWisdom Biopharma Co., Ltd. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: TWP-201-11
Record Dates: First submitted 2021-04-29; First posted 2021-05-07 (Actual); Last update posted 2021-07-19 (Actual); Status verified 2021-07

CONDITIONS: Infertility
MeSH Terms: conditions — Infertility

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- TWP-201 (Experimental)
  Interventions: Drug: TWP-201
- placebo (Placebo Comparator)
  Interventions: Drug: placebo

INTERVENTIONS:
Drug: TWP-201 — a single subcutaneous injection
  Arms: TWP-201
Drug: placebo — a single subcutaneous injection
  Arms: placebo

SUMMARY:
This study is a randomized, double-blind, placebo-controlled, single dose, escalation, phase I clinical trial to evaluate the safety and tolerability of recombinant human follicle stimulating hormone Fc fusion protein injection (TWP-201) in healthy female subjects. The objective of the trial is to evaluate the safety and tolerability of TWP-201 in healthy female subjects.

ELIGIBILITY:
Inclusion Criteria:

* Body weight ≥ 45 kg, 19 ≤ body mass index (BMI) ≤ 28 kg /m2;
* Women with sexual experience, potential fertility and regular menstrual cycle (25-34 days) (including boundary value);
* The levels of sex hormones were normal or abnormal without clinical significance at the time of screening;
* The physiological structure of uterus and bilateral ovaries was normal or abnormal by ultrasound examination, without clinical significance;

Exclusion Criteria:

* Known the history of stage III / IV endometriosis, submucosal myoma and endocrine abnormality within 6 months before enrollment;
* Known the history of ovarian hyperstimulation syndrome (OHSS);
* Premature ovarian failure, decreased ovarian reserve function (Antral Follicle Counting < 3), high ovarian response, polycystic ovary syndrome, unexplained vaginal bleeding or endometrial hyperplasia;
* Any FSH or HMG preparations were used within 3 months before the first study;
* Pregnancy or lactating women.

Ages: 18 Years to 42 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 48 (Estimated)
Dates: Start 2021-05-17 (Actual); Primary Completion 2022-10-31 (Estimated); Study Completion 2022-12-31 (Estimated)

PRIMARY OUTCOMES:
Incidence of adverse events, serious adverse and abnormal laboratory values event (defined by the Common Terminology Criteria for Adverse Events version 5.0 (CTCAE V5.0)). | An average of 1 year

SECONDARY OUTCOMES:
Maximum measured plasma concentration (Cmax) of TWP-201; | 28 days
Time to maximum plasma concentration (Tmax) of TWP-201; | 28 days
Half-life (T1/2) of TWP-201. | 28 days
Pharmacodynamics(PD). | 28 days
  Determination of serum concentrations of FSH, E2 and LH after dosing.
Pharmacodynamics(PD). | 28 days
  The number of follicles after dosing. The size of follicles after dosing.
Immunogenicity profile of TWP-201. | 28 days
  Blood samples will be collected from subjects post treatment for assessment to detect the presence of anti-drug antibodies and neutralizing antibodies.

CONTACTS AND LOCATIONS:
Overall Officials: Shengbin Ren, Principal Investigator — Medical Center
Locations (1):
- West China Second University Hospital, Sichuan University, Chengdu, Sichuan, China

IPD SHARING:
Plan to Share IPD: No